CLINICAL TRIAL: NCT01854515
Title: Comparison of Efficacy of Nebulizing Budesonide and Intravenous Dexamethasone Before Extubation on Prevention of Post-extubation Complications in Intensive Care Unit Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saeed Abbasi (Other)
Responsible Party: Sponsor-Investigator, Saeed Abbasi, Assistant Professor in Anesthesiology, Isfahan University of Medical Sciences
Organization: Isfahan University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 391387
Record Dates: First submitted 2013-05-13; First posted 2013-05-15 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Respiratory Sounds
MeSH Terms: conditions — Respiratory Sounds | interventions — Budesonide; dexamethasone acetate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Budesonide (Active Comparator): 1 mg diluted in 4 cc of sterile water for 20 minutes, one hour preceding extubation. After extubation patients received nebulizing Budesonide via oxygen mask at the same dose every 12 h. for 48 h.
  Interventions: Drug: Budesonide
- Dexamethasone (Experimental): 0.15 mg/kg before extubation. After extubation, the administration of intravenous Dexamethasone continued at the same dose every 12 h. for 48 h.
  Interventions: Drug: Dexamethasone acetate

INTERVENTIONS:
Drug: Budesonide
  Arms: Budesonide
Drug: Dexamethasone acetate
  Arms: Dexamethasone

SUMMARY:
The present study was aimed at investigating the efficacy of nebulizing Budesonide sin comparison with intravenous Dexamethasone before extubation in prevention of post-extubation complications amongst patients admitted in intensive care unit.

In this double-blind randomized clinical trial study, 90 patients (age between 18 to 65) who are intubated (at least for 48 hours) and now are ready for extubation will be enrolled in the study after obtaining a written informed consent from their parents or guardians.

The investigators divide our patients randomly into two equal groups.

-In the budesonide group patients underwent a therapy with nebulizing Budesonide at a dose of 1 mg diluted in 4 cc of sterile water for 20 minutes, one hour preceding extubation. After extubation patients received nebulizing budesonide via oxygen mask at the same dose every 12 hours for 48 h.i In dexamethasone group intravenous dexamethasone was administered to patient at a dose of 0.15 mg/kg before extubation. After extubation, the administration of intravenous Dexamethasone continued at the same dose every 12 h. for 48 h.

Another anesthesiologist who is unaware about kind of medication, will evaluate the patients for severity of stridor. We will record the vital sings and grade of stridor every 6 hour. Respiratory rate (RR), heart rate (HR), blood pressure (BP) and oxygen saturation (SPO2) were recorded for each patient immediately before aerosol administration (time 0) and at 30 and 60 min; and 2,4,8,12,24,36 and 48 hrs. After extubation then the presence of stridor (heard with the aid of stethoscope) was recorded within 48 hr of extubation

ELIGIBILITY:
Inclusion Criteria:

1. Patients' age 18-65 years old
2. Intubated for more than 48 hours after surgery
3. Met the weaning criteria defined as respiratory rate < 30 breaths / min, negative tidal volume > 5 ml/kg ideal body weight, and shallow index (respiratory rate/tidal volume) < 105 breaths / min/L

Exclusion Criteria:

1. Any history of corticosteroid therapy in previous week
2. Nasal or throat disease / surgery
3. Pulmonary airway disease
4. Gastrointestinal bleeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
post extubation stridor | After extubation until 48 hours
  Until 48 hours after extubation we documented if there is stridor in examination

CONTACTS AND LOCATIONS:
Locations (1):
- Alzahra University Hospital, Isfahan, Isfahan, Iran